CLINICAL TRIAL: NCT00668395
Title: Effects of CYP2B6 Genetic Polymorphisms on Efavirenz Pharmacokinetics, Autoinduction and Drug Interactions in Healthy Volunteers.
Brief Title: Effects of CYP2B6 Genetic Polymorphisms on Efavirenz Pharmacokinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1010002585 | 0704-14
Record Dates: First submitted 2007-11-27; First posted 2008-04-29 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: HIV
Keywords: CYP2B6; Efavirenz; Pharmacokinetics; Pharmacogenetics; Drug-Interactions
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CYP2B6*1/*1 genotype (Other): Efavirenz clearance in this genotype was compared with the other genotypes
  Interventions: Drug: Efavirenz
- CYP2B6*1/*6 (Other): Efavirenz clearance in this genotype was compared with the other genotypes
  Interventions: Drug: Efavirenz
- CYP2B6*6/*6 (Other): Efavirenz clearance in this genotype was compared with the other genotypes
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Efavirenz — The metabolism and pharmacokinetics of efavirenz were assessed at a single 600 mg oral dose of efavirenz and after subjects took multiple doses of efavirenz (600 mg/day orally for 17 days).
  Other Names: Sustiva

SUMMARY:
1. To see how the liver breaks down efavirenz by an enzyme called CYP2B6. It is suggested that when Efavirenz is taken repeatedly it may increase the amount of CYP2B6 in your liver and thus speed up your liver's ability to get rid of efavirenz from your body. This may render efavirenz and other medications ineffective.
2. To see how efavirenz interact with other drugs taken at the same time with it.
3. To see if genetic differences can change the way how the liver breaks down efavirenz and its interactions with other co-administered drugs.

DETAILED DESCRIPTION:
The human hepatic cytochrome P450 2B6 (CYP2B6) is a key enzyme in the metabolism of a growing list of clinically important drugs, environmental chemicals (e.g. toxicants and carcinogens) and endogenous substances. The expression and activity of this enzyme varies widely among individuals, probably due to genetic polymorphisms in the CYP2B6 gene and drug interactions. This variability, in turn, likely contributes to variable response to those drugs primarily metabolized by CYP2B6. In deed, several drugs that are substrates of CYP2B6 exhibit large pharmacokinetic differences among individuals and their use is associated with unpredictable drug interactions. Therefore, identifying mechanisms and factors that might influence CYP2B6 activity is important to the safe and effective use of its substrates. An important characteristic of several clinically important CYP2B6 substrate drugs that include efavirenz, nevirapine, cyclophosphamide, artemisinin and ifosfamide is their ability to enhance their own clearance upon repeated dosing, a process known as autoinduction of metabolism. Drugs that autoinduce metabolism also exhibit multiple interactions with drug metabolizing enzymes other than CYP2B6 (e.g. CYP3A, CYP2C9 and CYP2C19), and drug transporters (e.g. p-glycoprotein). As most of these medications are used in combination with other drugs, their potential to alter the pharmacokinetics of co-administered drugs is very high. We hypothesize that CYP2B6 genetic variants that influence constitutive CYP2B6 expression and activity contribute to interindividual variability in steady-state exposure of the autoinducer drugs and in the drug interactions that ensue. We will determine the impact of CYP2B6 genetic variants, typically the CYP2B6*6 allele, on the time-course and extent of autoinduction of metabolism and the consequences of differential autoinduction on drug interactions, using efavirenz (a known CYP2B6 substrate and an autoinducer) as a model drug. Thus, single (600 mg oral dose) and steady-state (600 mg/day) pharmacokinetics of efavirenz will be assessed in healthy subjects genotyped for the CYP2B6*6 allele. Trough concentrations of efavirenz and its metabolites will be collected during the course of efavirenz treatment. Efavirenz exposure will be compared between the genotypes after autoinduction. An autoinduction pharmacokinetic model will be developed to characterize the dynamics and time courses of autoinduction in the different genotypes. The potential impact of differences in efavirenz exposure on drug interactions will be determined by measuring the in vivo activity of selected CYP enzymes, using isoform specific substrate probes [omeprazole (CYP2C19), tolbutamide (CYP2C9), caffeine (CYP1A2) and midazolam (CYP3A)] at single and after multiple (steady-state) dosing with efavirenz.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 49 years old.
2. HIV negative. All potential subjects will be HIV tested at screening visit.
3. Healthy individuals without any significant medical condition.
4. Adherence to the study dietary restrictions.
5. Nonsmoker or individuals willing to refrain from smoking or use of tobacco or marijuana for at lest one month prior to and until the completion of the study. The entire study lasts for 30 days.
6. Ability to commit the time requested for this study.

Exclusion Criteria:

1. History or current HIV infection.
2. Life style that places you at a higher risk for contracting HIV (e.g. drug abuse, excessive alcohol drinking, and having multiple sexual partners).
3. Does not consent to HIV testing.
4. Underweight (weigh less than 52 kg or 114 lb) or overweight (body mass index (BMI) greater than 32).
5. History or current alcohol or drug abuse (more than 3 alcoholic drinks per day on a regular basis).
6. History of intolerance or allergic reaction (e.g. rash) to efavirenz, midazolam, tolbutamide, caffeine, or omeprazole.
7. History or current significant health conditions such as heart, liver, or kidney.
8. History or current psychiatric illness such as depression, anxiety, or nervousness.
9. History or current gastrointestinal disorders such as persistent diarrhea or malabsorption that would interfere with the absorption of orally administered drugs.
10. Individuals having a serious infection within the last month.
11. Donation of blood within the past two months.
12. Blood hemoglobin less than 12.5 mg/dl.
13. Individuals who are regularly taking prescriptions, over-the-counter, herbal or dietary supplements, alternative medications, or hormonal agents (i.e. oral contraceptives, intera-uterine device with hormones).
14. Females with a positive pregnancy test.
15. Breastfeeding.
16. Females of child-bearing potential who are unable or unwilling to either practice abstinence or use two non-hormonal forms of birth control (e.g. condom, contraceptive foams) up until the study completion, which will take a total of 30 days.
17. Participation in a research study or use of an investigational drug in the last two months.
18. An employee or student under supervision of any of the investigators of this study.
19. Individuals who cannot state a good understanding of this study including risks and requirements; are unable to follow the rules of this study.
20. Individuals with a gene type (DNA) that does not match one of the available genetic slot categories.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeruesenay Desta, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana Clinical Research Center (ICRC), Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana

REFERENCES:
- [Background] Turpeinen M, Raunio H, Pelkonen O. The functional role of CYP2B6 in human drug metabolism: substrates and inhibitors in vitro, in vivo and in silico. Curr Drug Metab. 2006 Oct;7(7):705-14. doi: 10.2174/138920006778520633. PMID 17073575
- [Background] Hodgson E, Rose RL. The importance of cytochrome P450 2B6 in the human metabolism of environmental chemicals. Pharmacol Ther. 2007 Feb;113(2):420-8. doi: 10.1016/j.pharmthera.2006.10.002. Epub 2006 Oct 24. PMID 17157385
- [Background] Ekins S, Wrighton SA. The role of CYP2B6 in human xenobiotic metabolism. Drug Metab Rev. 1999 Aug;31(3):719-54. doi: 10.1081/dmr-100101942. No abstract available. PMID 10461547
- [Background] Lang T, Klein K, Fischer J, Nussler AK, Neuhaus P, Hofmann U, Eichelbaum M, Schwab M, Zanger UM. Extensive genetic polymorphism in the human CYP2B6 gene with impact on expression and function in human liver. Pharmacogenetics. 2001 Jul;11(5):399-415. doi: 10.1097/00008571-200107000-00004. PMID 11470993
- [Background] Lang T, Klein K, Richter T, Zibat A, Kerb R, Eichelbaum M, Schwab M, Zanger UM. Multiple novel nonsynonymous CYP2B6 gene polymorphisms in Caucasians: demonstration of phenotypic null alleles. J Pharmacol Exp Ther. 2004 Oct;311(1):34-43. doi: 10.1124/jpet.104.068973. Epub 2004 Jun 9. PMID 15190123
- [Background] Klein K, Lang T, Saussele T, Barbosa-Sicard E, Schunck WH, Eichelbaum M, Schwab M, Zanger UM. Genetic variability of CYP2B6 in populations of African and Asian origin: allele frequencies, novel functional variants, and possible implications for anti-HIV therapy with efavirenz. Pharmacogenet Genomics. 2005 Dec;15(12):861-73. doi: 10.1097/01213011-200512000-00004. PMID 16272958
- [Derived] Collins KS, Aruldhas BW, Metzger IF, Lu JBL, Heathman MA, Quinney SK, Desta Z. A Population Pharmacokinetic Approach to Understand the Effect of Efavirenz on CYP3A Activity in Healthy Volunteers Using Midazolam as a Probe. CPT Pharmacometrics Syst Pharmacol. 2025 Dec;14(12):2095-2106. doi: 10.1002/psp4.70116. Epub 2025 Sep 24. PMID 40991845
- [Derived] Robarge JD, Metzger IF, Lu J, Thong N, Skaar TC, Desta Z, Bies RR. Population Pharmacokinetic Modeling To Estimate the Contributions of Genetic and Nongenetic Factors to Efavirenz Disposition. Antimicrob Agents Chemother. 2016 Dec 27;61(1):e01813-16. doi: 10.1128/AAC.01813-16. Print 2017 Jan. PMID 27799204
- [Derived] Metzger IF, Quigg TC, Epstein N, Aregbe AO, Thong N, Callaghan JT, Flockhart DA, Nguyen AT, Stevens CK, Gupta SK, Desta Z. Substantial effect of efavirenz monotherapy on bilirubin levels in healthy volunteers. Curr Ther Res Clin Exp. 2014 Sep 27;76:64-9. doi: 10.1016/j.curtheres.2014.05.002. eCollection 2014 Dec. PMID 25352936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects from self -referrals, campus fliers, Indiana University's Clinical Trials Webpage, community bulletin boards and newspaper were enrolled. All subjects were studied at the Indiana Clinical Research Center. Recruitment was completed within 3 years (8/20/07 to 4/15/10).
Pre-assignment Details: The study was initially designed to enroll subjects with prespecified CYP2B6 genotype (*1/*1, *1/*6, and *6/*6; n=20 each), but it was later modified in which subjects were enrolled without pregenotype information and genotype was performed post-hoc.
Groups:
- CYP2B6*1/*1 Genotype Group; CYP2B6*1/*6 Genotype Group; CYP2B6*6/*6 Genotype Group: 1. Efavirenz clearance following a single 600 mg oral dose of efavirenz and after multiple doses of efavirenz (600 mg/day orally for 17 days) was analyzed in normal metabolizer of CYP2B6 (CYP2B6*1/*1 genotype), intermediate metabolizer (CYP2B6*1/*6 genotype) and slow metabolizer (CYP2B6*6/*6).
     During the study, the design was slightly modified to sequentially enroll instead of allocation based on specific genotype, and genotype effect was analyzed post-hoc.
  2. The activities of CYP1A2, CYP2C9, CYP2C19, CYP3A were determined in all subjects (without regard to CYP2B6 genotype) using the metabolism of isoform selective probe substrates during the single dose (600 mg efavirenz orally) and after intake of multiple doses of efavirenz (600 mg/day efavirenz orally for 17 days) to assess efavirenz mediated drug interactions.
Period: Overall Study
Arm/Group | CYP2B6*1/*1 Genotype Group | CYP2B6*1/*6 Genotype Group | CYP2B6*6/*6 Genotype Group
Started | 45 | 22 | 6
Completed | 39 | 16 | 5
Not Completed | 6 | 6 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CYP2B6*1/*1: Normal metabolizer
- CYP2B6*1/*6: Intermediate metabolizer
- CYP2B6*6/*6: Slow metabolizer
- Total: Total of all reporting groups
Arm/Group | CYP2B6*1/*1 | CYP2B6*1/*6 | CYP2B6*6/*6 | Total
Number analyzed (Participants) | 45 | 22 | 6 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (10.2) | 29.5 (9.9) | 23.2 (3.9) | 28.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 6 | 4 | 27
  Male | 28 | 16 | 2 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 4 | 3 | 16
  White | 35 | 14 | 3 | 52
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] — A number of demographic parameters were collected at screening and during the completion of the study (exit).
  kg/m2 | 23.9 (3.5) | 25.4 (4.1) | 22.0 (3.0) | 24.2 (3.7)
Body weight [Mean (Standard Deviation); unit: kg] | 73.6 (13) | 77.2 (14.1) | 65 (5.3) | 74 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: Effect of CYP2B6 Genotype on Efavirenz Clearance
Description: Efavirenz clearance is a measure of rate of elimination of the drug from the body. We used this measure to evaluate differences in rate of elimination of efavirenz at a single dose and after multiple dosing within three CYP2B6 genotypes (CYP2B6*1/*1, *1/*6 and CYP2B6*6/*6). Efavirenz clearance was measured in normal metabolizer of CYP2B6 (CYP2B6*1/*1 genotype), intermediate metabolizer (CYP2B6*1/*6) and slow metabolizer (CYP2B6*6/*6) at a single 600 mg oral dose of efavirenz and then after multiple dosing (autoinduction), i.e., the administration of efavirenz (600 mg/day) for 17 days. Single and multiple dose efavirenz clearance was measured and compared to determine the extent of autoinduction within this genotype group.
Time Frame: Efavirenz clearance at single dose and multiple dose stratified by CYP2B6 genotypes
Measure: Mean (Standard Deviation); unit: ml/h/kg
Arm/Group | CYP2B6*1/*1 | CYP2B6*1/*6 | CYP2B6*6/*6
Number analyzed (Participants) | 38 | 17 | 5
ml/h/kg
  Single efavirenz dose | 93.35 (21.74) | 76.08 (21.59) | 51.03 (12.06)
  Multiple efavirenz dose | 50.05 (36.04) | 119.90 (39.15) | 80.12 (38.12)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study period which was approximately 30 days. I some case, follow-up assessment was carried out up to 2 months after completion of the study and subject was discharged from the study.
Arm/Group | CYP2B6*1/*1 | CYP2B6*1/*6 | CYP2B6*6/*6
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/22 | 0/6
Other Adverse Events (participants affected / at risk) | 0/45 | 0/22 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No